CLINICAL TRIAL: NCT04759274
Title: Diuretic Tuner Clinical Decision Support Mobile Device Application for Diuretic Titration in Hypervolemic States
Brief Title: Diuretic Tuner Clinical Decision Support
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kamalanathan Sambandam, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2020-1124
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Edema; Hypervolemia; Chronic Kidney Diseases; Nephrotic Syndrome
MeSH Terms: conditions — Edema; Renal Insufficiency, Chronic; Nephrotic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Diuretic Tuner users (Experimental): The Diuretic Tuner is a mobile device application that integrates a patient's estimated dry weight and starting diuretic dose (both defined by a healthcare provider) with daily weights and blood pressures to provide individualized guidance to the patient in day-to-day adjustments to his or her diuretic regimen. In addition, the application generates a diary of daily weights, blood pressures, fluid intake, and medication compliance.
  Interventions: Device: Diuretic Tuner

INTERVENTIONS:
Device: Diuretic Tuner — Mobile device application for diuretic dose titration

SUMMARY:
This purpose of this study is to determine the effectiveness of a mobile phone application in helping to control body swelling in patients with kidney problems. The application will help in the day to day adjustments in diuretic medication dosing.

Participants in this study will have an application loaded on to their mobile phone by the study team and be taught how to use it over a 2 hour visit. Participants will need to check their blood pressure and weight daily and enter this information into the mobile phone application every day. Participants will need to follow daily instructions in their medication dosing provided by the application. There will be periodic blood testing. This will happen at 2 weeks, 90 days, and up to 4 other times if necessary. At the end of the study there is a 2 hour study visit during which participants will answer a survey. The total length of the study is 90 days.

DETAILED DESCRIPTION:
Study Population: 30 subjects with signs of hypervolemia and either nephrotic syndrome or chronic kidney disease 4 to 5.

Study Intervention: This is a nonrandomized, uncontrolled trial. The Diuretic Tuner mobile device application will be deployed in the care of hypervolemic subjects as defined in the study population. The Diuretic Tuner will integrate each subject's estimated dry weight and starting diuretic dose (both defined by healthcare provider) with daily weights and blood pressures to provide individualized guidance to the subject in day-to-day adjustments to his or her diuretic regimen. In addition, the application will generate a diary of daily weights, blood pressures, fluid intake, and medication compliance. There will be no control arm as this first phase is to test feasibility/safety.

Study Outcome Measures: The primary outcomes of interest will focus on the achievement of the provider-defined estimated dry weight (both the time to achieving this target as well as the subsequent stability in weights around this target). Secondary outcomes of interest include safety metrics (3-month hospitalization rates, rates of hypokalemia, and rates of acute kidney injury) and tool usability (assessed through surveys evaluating ease of comprehension and satisfaction).

ELIGIBILITY:
Inclusion Criteria:

* The presence of nephrotic range proteinuria (> 3 g/d proteinuria by 24hr urine protein, 24hr urine albumin, spot urine protein/creatinine ratio, or spot urine albumin/creatinine ratio) or stage 4 or 5 chronic kidney disease (estimated glomerular filtration rate < 30 mL/min/1.73 m2 by Modification of Diet in Renal Disease equation) PLUS
* Clinical signs of hypervolemia present (lower extremity edema, ascites, or pleural effusions) with an estimated dry weight (defined as edema-free weight without orthostatic hypotension) 5 lbs less than enrollment body weight

Exclusion Criteria:

* Weight < 100 lbs or > 300 lbs.
* Autonomic insufficiency resulting in orthostatic hypotension at screening
* Hypokalemia at enrollment (defined as serum potassium < 3.5 mmol/L)
* Moderate to severe hyponatremia at enrollment (defined as serum sodium < 130 mmol/L)
* Serum creatinine > 6 mg/dL or > 1.5 times baseline
* Patients who are unable or unwilling to measure their home blood pressures and weights
* Patients without a working phone number and smart phone device
* Expectation that the patient will require dialysis initiation within < 3 months
* Expected lifespan of < 6 months
* The presence of a medical condition that would interfere with effectively using the Diuretic Tuner (dementia, illiteracy, or blindness)
* Pregnant patients
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Mean time to the attainment of dry weight | 90 days
  Mean time in days to the attainment of the provider-specified estimated dry weight
90 day weight variability | 90 days
  90 day weight variability around the target dry weight, as assessed by standard deviation

SECONDARY OUTCOMES:
Composite rate of hospitalization, hypokalemia, or acute renal insufficiency | 90 days
  90 day adverse event rate for the composite outcome including hospitalization for volume-related complications (hypervolemia, hypovolemia, or electrolyte disturbance), hypokalemia (serum potassium < 3.5 mmol/L), or acute renal insufficiency (serum creatinine ≥ 2 times baseline or > 6 mg/dL)
Diuretic Tuner usability assessed by user survey | 90 days
  Diuretic tuner usability (measured by Likert scale survey administered to each subject at the end of 90 days)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No